CLINICAL TRIAL: NCT05108272
Title: Comparison of Cosmetic and Functional Outcome of Silicone Sheeting and Micro-needling on Hypertrophic Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2021/2
Record Dates: First submitted 2021-08-17; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silicone Sheeting (Active Comparator): After explaining and taking consent from the patient about the intervention, pre intervention assessment will be made. Silicone gel sheet (Rystoraº) will be used at scar wound for 16 hours every day for 3 months. After 3 months post intervention assessment will be made.
  Interventions: Procedure: Percutaneous Collagen Induction
- Microneedling (Experimental): After explaining and taking consent from the patient about the intervention, pre- intervention assessment will be made. Derma pen (Dr.Pen auto Microneedle system Ultima-A6) with 36 needles per cm2 will be used with adjustable depth of 0.5mm to 2mm. Micro-needling will be performed in 3 axis,1st in vertical, then horizontal and then oblique direction to the point of uniform petechial bleed. Four sessions at 3 weekly intervals will be performed. Final assessment will be made after 3 months of first intervention
  Interventions: Procedure: Microneedling

INTERVENTIONS:
Procedure: Microneedling — Derma Pen is an electric device, used for microneedling. Derma pen has a Cartridge which has microneedles fitted. These needles penetrate the skin upto 2mm
  Other Names: Percutaneous Induction
  Arms: Microneedling
Procedure: Percutaneous Collagen Induction — It is self-adhesive sheet made from medical graded Silicone. It has micropore technology which entraps moisture where it is needed on scared skin.
  Arms: Silicone Sheeting

SUMMARY:
Hypertrophic scars and keloids are frequently encountered in plastic surgery OPD. due to any reason, the normal wound healing is impaired, hypertrophic scars or keloids occur. These are thickened, wide and raised scars. Many treatment options are presented over time, but most of the treatments remain insufficient. Treatment options include massage therapy, silicone sheet, occlusive dressings, pressure garments, adhesive tape, intra-lesional steroid injections, laser therapy, cryotherapy, radiotherapy, 5-fluorouracil, interferons, bleomycin, imiquimod 5%cream, tranilast, botulin toxin and surgical excision. In this Study outcomes of treatment with silicone sheeting and microneedling will be compaired.

DETAILED DESCRIPTION:
Hypertrophic scars and keloids are one of difficult conditions to treat. Prevention of abnormal scaring is more effective than treatment, so avoiding unnecessary wounds in patients is a solution but flawed one. Many treatment options are presented over time, but most of the treatments remain insufficient. Treatment options include massage therapy, silicone sheet, occlusive dressings, pressure garments, adhesive tape, intra-lesional steroid injections, laser therapy, cryotherapy, radiotherapy, 5-fluorouracil, interferons, bleomycin, imiquimod 5%cream, tranilast, botulin toxin and surgical excision. Silicone sheeting is considered first line therapy of hypertrophic scar. It works by maintaining hydration and occlusion at scar site. But silicone sheeting is expensive and need 12 to 24 hours of constant application daily for at least 2 months for desired results. Level 1, 2 and 3 evidences show newer technique 'percutaneous collagen induction(micro-needling)', shows significant improvement in hypertrophic scars. Micro-needling causes controlled dermal injury to initiate inflammatory and healing reaction, which in turn leads to remodelling of collagen and stimulate regeneration of scared skin. Silicone sheets is an expensive treatment requiring multiple applications and are often difficult to use in hot and humid environment. These reasons often lead to poor patient compliance. Keeping these issues in mind we planned to study an alternative option i.e. micro-needling, which is relatively of low cost and better patient acceptability. When doing the literature review the investigator found scanty evidence so the investigator decided to perform this RCT.

ELIGIBILITY:
1. All the patients presenting with hypertrophic scars ≥1cm in size
2. Any age
3. Both genders

Exclusion criteria:

1. Pregnant or lactating mothers
2. Patients who already taking systemic steroid as confirmed through clinical record
3. Patients with renal failure or liver failure as confirmed through clinical history
4. Patient with uncontrolled diabetes.
5. Patients who received treatment for keloids or hypertrophic scar in past.
6. Patients with active inflammation in area of hypertrophic scar or in its vicinity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Cosmetic Outcome | 3 Months
  It will be assessed using, Vancouver scar scale at time of presentation and at 3 months after the intervention. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented. Vancouver Scar Scale is a 13 points scale and includes four parameters, pigmentation, vascularity pliability and height of scar.13 It is an objective scale and examining doctor will assess and record score out of 13. Lesser the score better is the scar.

SECONDARY OUTCOMES:
Itching at scar site | 3 Months
  It will be assessed at the time of presentation and at 3 months after the intervention using severity of pruritus scale. It is 4 point rating scale from 0 (no itch) to 3(severe itch disturbing the sleep) assessing severity of pruritus within 24-hours recall period. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented.
Pain At scar Site | 3 Months
  Patient will be asked to rate his/her current, best and worst pain level over past 24 hours on scale of 0 (no pain) to 10 (worst pain imaginable). Pain at scar site will be assessed at time of presentation and then at 3 months after start of the treatment. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented. This scale is chosen due to its high feasibility and good compliance.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Foundation University Islamabad, Islamabad, Federal
  - FFH, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No